CLINICAL TRIAL: NCT01907555
Title: Clinical, Molecular and Physiopathological Study of Cohen Syndrome and Cohen-like Syndromes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE PHRC N 2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Cohen Syndrome
MeSH Terms: conditions — Cohen syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- - Patients presenting Cohen syndrome and two VPS13B mutations
- Patients presenting Cohen syndrome without a VPS13B mutation
- Patients presenting neutropenia

SUMMARY:
This project will make it possible to better understand the natural history of Cohen Syndrom and the phenotypes associated with mutations in the VPS13B gene, to improve the therapeutic management of patients. It will also provide a better description of Cohen-like syndrome for genetic counselling for the families concerned.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Cohen syndrome and two VPS13B mutations
* who accept a clinical evaluation, and to provide at least one blood sample
* Patients presenting the diagnostic criteria of Cohen syndrome, but without a VPS13B mutation
* Patients presenting neutropenia or pigmentary retinopathy and at least one of the following signs, after exclusion of any other syndrome: mental retardation, microcephaly, truncal obesity

Exclusion Criteria:

* - Patients who do not meet the clinical and/or molecular criteria
* Patients who do not wish to provide a blood sample for question 1,
* Patients who have not provided written informed consent,
* Pregnant or breast-feeding women,
* Persons not covered by National Health Insurance and persons under guardianship or in prison.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohen syndrome
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07-24 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
spectrum of mutations VPS13B | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France